CLINICAL TRIAL: NCT02548650
Title: Pharmacodynamic Effects of Vorapaxar as an Add-On Antiplatelet Therapy in Patients With and Without Diabetes Mellitus: The Optimizing Anti-Platelet Therapy In Diabetes MellitUS (OPTIMUS)-5 Study
Brief Title: Vorapaxar as an Add-On Antiplatelet Therapy in Patients With and Without Diabetes Mellitus
Acronym: OPTIMUS-5
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIS 53377
Record Dates: First submitted 2015-09-08; First posted 2015-09-14 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-01

CONDITIONS: Myocardial Infarction; Diabetes Mellitus; Peripheral Arterial Disease
Keywords: myocardial infarction; diabetes mellitus; vorapaxar; peripheral arterial disease
MeSH Terms: conditions — Myocardial Infarction; Diabetes Mellitus; Peripheral Arterial Disease | interventions — vorapaxar; Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patients with diabetes (Experimental): Triple therapy (vorapaxar 2.5mg od plus clopidogrel 75 mg od and aspirin 81 mg od) will be administered for 30 days; then patients will stop aspirin and will take dual treatment (vorapaxar 2.5mg od plus clopidogrel 75 mg od ) for other 30 days.
  Interventions: Drug: Vorapaxar; Drug: Clopidogrel; Drug: Aspirin
- Patients without diabetes (Active Comparator): Triple therapy (vorapaxar 2.5mg od plus clopidogrel 75 mg od and aspirin 81 mg od) will be administered for 30 days; then patients will stop aspirin and will take dual treatment (vorapaxar 2.5mg od plus clopidogrel 75 mg od ) for other 30 days.
  Interventions: Drug: Vorapaxar; Drug: Clopidogrel; Drug: Aspirin

INTERVENTIONS:
Drug: Vorapaxar — Triple therapy with DAPT plus vorapaxar (vorapaxar 2.5mg od plus clopidogrel 75 mg od and aspirin 81 mg od) will be administered for 30 days; then patients will stop aspirin and will take dual treatment (vorapaxar 2.5mg od plus clopidogrel 75 mg od ) for other 30 days
  Other Names: Zontivity
Drug: Clopidogrel — Triple therapy with DAPT plus vorapaxar (vorapaxar 2.5mg od plus clopidogrel 75 mg od and aspirin 81 mg od) will be administered for 30 days; then patients will stop aspirin and will take dual treatment (vorapaxar 2.5mg od plus clopidogrel 75 mg od ) for other 30 days
  Other Names: Plavix
Drug: Aspirin — Triple therapy with DAPT plus vorapaxar(vorapaxar 2.5mg od plus clopidogrel 75 mg od and aspirin 81 mg od) will be administered for 30 days; then patients will stop aspirin and will take dual treatment (vorapaxar 2.5mg od plus clopidogrel 75 mg od ) for other 30 days
  Other Names: ASA

SUMMARY:
Dual antiplatelet therapy (DAPT) with aspirin and a P2Y12 receptor inhibitor, more frequently clopidogrel, represents the standard of care for the long-term secondary prevention of atherothrombotic events in patients with myocardial infarction (MI) or peripheral arterial disease (PAD). However, rates of ischemic recurrences remain high. Vorapaxar is a protease-activated receptor (PAR)-1 inhibitor, which exerts potent inhibition of thrombin-mediated platelet aggregation. Patients with diabetes mellitus (DM) are known to be at increased risk of recurrent atherothrombotic events, which translates into worse outcomes, despite the use of standard of care therapy. This is in part due to the hyperreactive platelet phenotype, which characterizes DM patients, and to inadequate response to oral antiplatelet agents, including clopidogrel. Therefore, vorapaxar is an attractive treatment option for DM patients with a prior MI. The pharmacodynamic (PD) effects of vorapaxar in DM patients and how these may differentiate from non-DM patients has not been explored. Further, the role of vorapaxar as part of a dual antithrombotic treatment regimen combined with clopidogrel (and stopping aspirin) represents another important area of clinical interest. The proposed prospective, parallel-design study conducted in patients post-MI or with PAD with and without DM will aim the assess the pharmacodynamic effects of vorapaxar in addition to standard DAPT with aspirin and clopidogrel as well as in combination with clopidogrel only following aspirin withdrawal.

DETAILED DESCRIPTION:
Dual antiplatelet therapy (DAPT) with aspirin and a P2Y12 receptor inhibitor, more frequently clopidogrel, represents the standard of care for the long-term secondary prevention of atherothrombotic events in patients with myocardial infarction (MI) or peripheral arterial disease (PAD). However, rates of ischemic recurrences remain high, in part due to the fact that other platelet signaling pathways, such as thrombin-induced platelet aggregation, continue to be activated. Vorapaxar is a novel, orally active, competitive and slowly reversible protease-activated receptor (PAR)-1 inhibitor, which exerts potent inhibition of thrombin-mediated platelet aggregation. It is approved for clinical use by the Food and Drug Administration for the reduction of thrombotic cardiovascular events in patients with a history of MI or with peripheral arterial disease. Patients with DM are known to be at increased risk of recurrent atherothrombotic events, which translates into worse outcomes, despite the use of standard of care therapy. This is in part due to the hyperreactive platelet phenotype, which characterizes DM patients, and to inadequate response to oral antiplatelet agents, including clopidogrel. Importantly, in DM patients with prior MI included in the TRA 2P trial, vorapaxar reduced the primary composite end point at 3 years by 27% and led to a greater absolute risk reduction compared with those without DM. Therefore, vorapaxar is an attractive treatment option for DM patients with a prior MI. However, to date the PD effects of vorapaxar in DM patients and how these may differentiate from non-DM patients has not been explored. Further, current trends in clinical practice are seeing many patients discontinue aspirin and maintain clopidogrel. Hence, the role of vorapaxar as part of a dual antithrombotic treatment regimen combined with clopidogrel (and stopping aspirin) represents another important area of clinical interest, in order to maximize ischemic protection while reducing the risk of bleeding. The proposed prospective, parallel-design study conducted in patients post-MI or with PAD with and without DM will aim the assess the pharmacodynamic effects of vorapaxar in addition to standard DAPT with aspirin and clopidogrel as well as in combination with clopidogrel only following aspirin withdrawal. Pharmacodynamic assessments will be performed at multiple time point, with different assays exploring multiple pathways of platelet aggregation.

ELIGIBILITY:
Inclusion criteria:

1. Patients with a prior MI between 2 weeks and 24 months or with PAD.
2. On DAPT with low-dose aspirin (81mg od) and clopidogrel (75mg od) as per standard-of-care for at least 14 days.
3. Age ≥ 18 years old.

Exclusion criteria:

1. History of acute coronary syndrome in the previous 2 weeks.
2. History of stroke, transient ischemic attack, or intracranial hemorrhage.
3. Active pathological bleeding, history of bleeding events or increased risk of bleeding.
4. Known severe hepatic impairment.
5. Use of strong cytochrome P450 3A4 inhibitors (e.g., ketoconazole, itraconazole, posaconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, boceprevir, telaprevir, telithromycin and conivaptan) or inducers (e.g., rifampin, carbamazepine, St. John's Wort and phenytoin).
6. On treatment with any oral anticoagulant (vitamin K antagonists, dabigatran, rivaroxaban, apixaban, edoxaban).
7. On treatment with any antiplatelet agent other than aspirin and clopidogrel in the past 14 days.
8. Creatinine clearance <30 mL/minute.
9. Platelet count <80x106/mL
10. Hemoglobin <10g/dL
11. Hemodynamic instability
12. Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-03-25 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Angiolillo, MD, PhD, Principal Investigator — University of Florida College of Medicine-Jacksonville
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franchi F, Rollini F, Kairouz V, Rivas Rios J, Rivas A, Agarwal M, Briceno M, Wali M, Nawaz A, Silva G, Shaikh Z, Maaliki N, Been L, Piraino J, Pineda AM, Suryadevara S, Soffer D, Zenni MM, Jennings LK, Bass TA, Angiolillo DJ. Pharmacodynamic Effects of Vorapaxar in Patients With and Without Diabetes Mellitus: Results of the OPTIMUS-5 Study. JACC Basic Transl Sci. 2019 Sep 1;4(7):763-775. doi: 10.1016/j.jacbts.2019.07.011. eCollection 2019 Nov. PMID 31998847

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Between March 2016 and October 2018, 71 patients agreed to participate in the study; 5 patients were not eligible for randomization due to the presence of an exclusion criteria. 66 patients (DM, n=30; non-DM, n=36) were exposed to at least one dose of study medication, representing the safety population.
Period: Triple Therapy
Arm/Group | Patients With Diabetes | Patients Without Diabetes
Started | 30 | 36
Completed | 29 | 32
Not Completed | 1 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4
Period: Double Therapy
Arm/Group | Patients With Diabetes | Patients Without Diabetes
Started | 29 | 32
Completed | 28 | 30
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Two patients were not compliant with medications and therefore excluded from the PD analysis. Thus, a total of 64 patients (DM, n=30; non-DM, n=34) represented the PD population of the study and were analyzed for baseline characteristics and PD data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With Diabetes | Patients Without Diabetes | Total
Number analyzed (Participants) | 30 | 34 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (8) | 56 (9) | 58 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 23 | 23 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 11 | 25
  White | 15 | 22 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
chronic kidney disease [Count of Participants; unit: Participants] | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximal Platelet Aggregation in DM
Description: Comparison of maximal platelet aggregation (%) measured by light transmittance aggregometry between between triple (vorapaxar plus DAPT) and dual (vorapaxar plus clopidogrel) therapy in diabetic patients
Time Frame: 30 days
Population: The PD population included all patients with PD data and without a major protocol deviation thought to affect the PD effects of vorapaxar, aspirin and clopidogrel. Two patients were not compliant with medications and therefore excluded from the PD analysis. Some patients did not have primary end point data but were considered for other analyses.
Measure: Mean (Standard Deviation); unit: percentage of aggregation
Groups:
- Triple Therapy: vorapaxar plus DAPT
- Dual Therapy: (vorapaxar plus clopidogrel)
Arm/Group | Triple Therapy | Dual Therapy
Number analyzed (Participants) | 30 | 30
percentage of aggregation | 65 (20) | 78 (20)
Statistical Analysis 1: Comparison: Triple Therapy vs Dual Therapy; The primary end point of our study was the comparison of CAT-induced MPA measured by LTA between triple (vorapaxar plus DAPT) and dual (vorapaxar plus clopidogrel) therapy. We hypothesized that dual therapy would be non-inferior to triple therapy after 30±5 days of treatment; Test type: Non-Inferiority — Under the null hypothesis that the mean aggregation between dual and triple therapy is not equal to 0 and a common standard deviation of 13%, a sample size of 28 patients per group with a valid primary end point time point allowed for the 95% confidence interval (CI) to stay within ± 10% with a 80% power and a two-sided alpha=0.05; p > 0.05, ANOVA; Mean Difference (Net) = 12, 95% CI 2-sided [3 to 21]

2. Secondary Outcome: Maximal Platelet Aggregation in Non-DM
Description: Comparison of maximal platelet aggregation (%) measured by light transmittance aggregometry between between triple (vorapaxar plus DAPT) and dual (vorapaxar plus clopidogrel) therapy in non-diabetic patients
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: percentage of aggregation
Arm/Group | Triple Therapy | Dual Therapy
Number analyzed (Participants) | 34 | 34
percentage of aggregation | 60 (15) | 70 (20)

ADVERSE EVENTS:
Time Frame: Study duration (60 days)
Arm/Group | Patients With Diabetes | Patients Without Diabetes
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/36
Other Adverse Events (participants affected / at risk) | 2/30 | 2/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Diabetes (N=30) | Patients Without Diabetes (N=36)
minor bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — hematuria
Chest pain (Cardiac disorders) | 1 (1) | 2 (2) — chest pain not requiring intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT02548650/Prot_SAP_000.pdf